CLINICAL TRIAL: NCT04576793
Title: Longitudinal Imaging of Microglial Activation in Different Clinical Variants of Alzheimer's Disease
Acronym: ADVISe
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Patrick Lao (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Patrick Lao, Associate Professor of Neurology, Columbia University
Organization: Columbia University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAS7810; R01AG063888 (NIH)
Record Dates: First submitted 2020-09-29; First posted 2020-10-06 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease
Keywords: Inflammation; PET scans; Cognitive Impairment; Posterior Cortical Atrophy; Logopenic Variant Primary Progressive Aphasia; Amnestic Alzheimer's Disease; MK-6240; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Inflammation; Cognitive Dysfunction | interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene; Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cognitive impairment (Experimental): * Mild Cognitive Impairment
  * Posterior cortical atrophy - a version of Alzheimer's disease with vision difficulties
  * Logopenic variant primary progressive aphasia - a version of Alzheimer's disease with language difficulties
  * Amnestic Alzheimer's disease - a "typical" version of Alzheimer's disease with memory difficulties
  Interventions: Drug: 11C-ER176; Drug: 18F-MK6240; Drug: 18F-Florbetaben; Procedure: Lumbar Puncture
- No cognitive impairment (Active Comparator): Healthy controls
  Interventions: Drug: 11C-ER176; Drug: 18F-MK6240; Drug: 18F-Florbetaben; Procedure: Lumbar Puncture

INTERVENTIONS:
Drug: 11C-ER176 — 11C-ER176 sticks to parts of the brain where there is inflammation. Past studies have shown that inflammation is present in the brains of patients with Alzheimer's disease. The purpose of this study is to determine if 11C-ER176 is able to accurately measure inflammation in patients with Alzheimer's disease. 11C-ER176 will be administered at activity up to 20 millicurie (mCi) per injection.
  Other Names: [11C] ER176
Drug: 18F-MK6240 — MK-6240 measures a protein called in the brain. MK-6240 is experimental but has been used in several human studies before and has been proven to accurately measure tau in the brain.
  Other Names: [18F-MK6240]
Drug: 18F-Florbetaben — Florbetaben has been approved by the FDA to help diagnose Alzheimer's disease. florbetaben measures amyloid in the brain.
  Other Names: [18F] Florbetaben
Procedure: Lumbar Puncture — Inflammation can also be measured by looking at certain proteins in the spinal fluid. In order to measure these proteins in the spinal fluid, the investigators will perform a lumbar puncture (spinal tap).
  Other Names: Spinal Tap

SUMMARY:
The purpose of this study is to determine how inflammation is related to other changes in the brain that occur during the progression of Alzheimer's disease. The investigators are also studying how inflammation is related to the symptoms that first occur in patients with Alzheimer's disease (AD). For this reason, the investigators are asking people with different versions of Alzheimer's disease and/or other related dementias to participate. This includes patients with:

* Mild Cognitive Impairment
* Posterior cortical atrophy - a version of Alzheimer's disease with vision difficulties
* Logopenic variant primary progressive aphasia - a version of Alzheimer's disease with language difficulties
* Amnestic Alzheimer's disease - a "typical" version of Alzheimer's disease with memory difficulties
* The investigators are also enrolling older adults with normal visual, language, and memory function.

DETAILED DESCRIPTION:
This study is being done to learn about inflammation in Alzheimer's disease so that the investigators can find out new ways to treat patients with this disease. Because Alzheimer's disease usually causes slow changes to the brain over time, in this study the investigators are going to perform different tests and then repeat some of them two years later.

Inflammation can be measured using a type of brain scan called a positron emission tomography (PET) scan. A PET scan uses very small amounts of a radioactive drug that is injected into a vein to create a special picture of the brain. The inflammation PET scan uses a drug called ER176. ER176 is an experimental drug but has been used in several human studies before. Once in the body, ER176 sticks to areas with lots of inflammation, and the PET scan allows us to see these areas.

Inflammation can also be measured by looking at certain proteins in the spinal fluid. In order to measure these proteins in the spinal fluid, the investigators need to perform a lumbar puncture (spinal tap). Certain genes that inherited from parents influence the amount of inflammation in the body. The investigators can study how genes affect inflammation in Alzheimer's disease by looking doing genetic tests on blood that collected from the vein.

The investigators can study how genes affect inflammation in Alzheimer's disease by doing genetic tests on blood. The investigators will also be testing blood for severe acute respiratory syndrome (SARS)- CoV-2 (the virus that causes COVID-19) antibodies. The investigators want to see if exposure to the virus that causes COVID-19 changes the amount of inflammation in the brain or not.

Along with inflammation, Alzheimer's disease is also associated with the build up of the proteins amyloid and tau in the brain. The investigators can measure these proteins using PET scans. The amyloid PET scan uses a drug called florbetaben that has been approved by the FDA to help diagnose Alzheimer's disease. The tau PET scan uses a drug called MK-6240. Like ER176, MK-6240 is experimental but has been used in several human studies before.

A brain MRI creates a high resolution picture of the brain. The brain MRI helps the investigators get more information from the PET scans, and can also tell the investigators the size and appearance of different brain structures. When someone has Alzheimer's disease, some of these brain structures get smaller or have altered appearance on MRI.

ELIGIBILITY:
Inclusion criteria:

1. Age 50 and over at time of screening.
2. At screening, must have no cognitive impairment, or meet criteria for amnestic Alzheimer's disease, posterior cortical atrophy, or logopenic variant primary progressive aphasia. Diagnoses will be made based on history, exam, neuropsychological testing, brain MRI, and consensus diagnosis.
3. Patients must have Clinical Dementia Rating scale score of 0.5 or 1 at enrollment. Controls must have Clinical Dementia Rating scale score of 0 at enrollment.
4. Subjects unable to provide informed consent must have a surrogate decision maker.
5. Written and oral fluency in English or Spanish.
6. Able to participate in all scheduled evaluations and to complete all required tests and procedures.
7. In the opinion of the PI, the subject must be considered likely to comply with the study protocol and to have a high probability of completing the study.

Exclusion criteria:

1. Past or present history of a brain disorder other than Alzheimer's disease (including presence of cortical infarct on MRI even in absence of clinical stroke).
2. Serious medical conditions, which make study procedures of the current study unsafe. Such serious medical conditions include uncontrolled epilepsy and multiple serious injuries.
3. Contraindication to MRI scanning.
4. Conditions precluding entry into the scanners (e.g. morbid obesity, claustrophobia, etc.).
5. Exposure to research related radiation in the past year that, when combined with this study, would place subjects above the allowable limits.
6. Exact medication exclusions are up to the discretion of the PI in consultation with the MD liaison.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-11-17 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
11C-ER176 Standardized Uptake Value Ratio | Up to 24 months
  The standardize uptake value ratio is the concentration of radioactivity measured from the 11C-ER176 PET scan in the cortex compared to the uptake in the cerebellum (pseudo-reference region).
18F-MK6240 Standardized Uptake Value Ratio | Up to 24 months
  The standardize uptake value ratio is the concentration of radioactivity measured from the 18F-MK6240 PET scan in the cortex compared to the uptake in the cerebellum (pseudo-reference region).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J. Lao, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available upon reasonable request from a qualified investigator.
Time Frame: Up to two weeks after review and approval of request.
Access Criteria: Investigator qualifications and previous work will be reviewed by PI. Subsequent email correspondence will relay technical criteria needed for access.